CLINICAL TRIAL: NCT02421822
Title: BMI Study for Children Ages 6-9 Years and Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ann McGaffey, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO14080265
Record Dates: First submitted 2015-03-26; First posted 2015-04-21 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fitwits Intervention (Experimental): Fitwits office tool and games
  Interventions: Other: Fitwits office tool and games

INTERVENTIONS:
Other: Fitwits office tool and games — Physician-led narration of Fitwits office tool during well child and subsequent visits over one year with distribution of Fitwits games during first visit.

SUMMARY:
The purpose of this study is to test the Fitwits office tool and games with 6-9 year old children and their parents to: 1) assist parent-child dyad with correct BMI status identification and understanding; 2) address nutrition, portion size, and activity cues; and, 3) track BMI trajectory over 12-month period.

DETAILED DESCRIPTION:
The investigators will study parents' perceptions of their child's BMI before and after the Fitwits intervention with a primary goal of improving parents' ability to identify their child's actual BMI status (underweight, healthy weight, overweight, or obese). Secondary goals are to measure changes in behaviors and BMI trajectories with repetitive use of the Fitwits office tool.

The study design is a longitudinal non-randomized intervention study with four time points (baseline, 3, 6, and 12 months). The investigators will recruit family medicine residents, fellows, and faculty at the investigators' three family health centers and enroll 150 parent/guardians and children aged 6-9 years at well child visits, regardless of initial BMI.

The investigators will use electronic health record-generated BMI percentages, the physician-led Fitwits Office Tool as the intervention, and self-reported surveys for the parent-child dyad. Surveys will record the BMI understanding -pre- and post-Fitwits intervention at each visit.

The investigators will compare the intervention to a control group residency-based family health center with usual care for child/parent dyads presenting at well child care and 12 months later. At this site the investigators will survey for correct parent identification of the child's BMI category.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-9 regardless of BMI status

Exclusion Criteria:

* non-English-speaking

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 487 (Actual)
Dates: Start 2015-06-14 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Improved parent correct identification of child BMI category (surveys) | one year
  improved correctness of BMI category selection on surveys over one year

CONTACTS AND LOCATIONS:
Overall Officials: Ann L McGaffey, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC St.Margaret Bloomfield/Garfield Family Health Center, Pittsburgh, Pennsylvania, United States